CLINICAL TRIAL: NCT01760915
Title: Severe Asthma Research Program (SARP) - University of Wisconsin
Brief Title: University of Wisconsin Severe Asthma Research Program III
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Washington University School of Medicine (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2012-0571; 4U10HL109168 (NIH); A534285 (Other: UW, Madison); R01HL115118 (NIH); MRTG-02-15-2022 (Other Grant/Funding Number: Foundation for Anesthesia Education and Research)
Record Dates: First submitted 2012-12-26; First posted 2013-01-04 (Estimated); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Asthma
Keywords: asthma; severe
MeSH Terms: conditions — Asthma; Lymphoma, Follicular | interventions — Helium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, DNA, RNA, sputum, urine, bronchial tissue, bronchoalveolar lavage, bronchial brushings, exhaled breath condensate
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Severe asthma: Subjects with severe asthma (SARP protocol definition)
  Interventions: Other: NC100182 Hyperpolarized 3He
- Well controlled asthma: Subjects with well controlled asthma
  Interventions: Other: NC100182 Hyperpolarized 3He
- Normal control: Subjects that are healthy normals
  Interventions: Other: NC100182 Hyperpolarized 3He

INTERVENTIONS:
Other: NC100182 Hyperpolarized 3He — Magnetic Resonance Imaging (MRI) will take place and include inhalation of hyperpolarized helium to construct an image of the lungs.
  Other Names: helium

SUMMARY:
The overall goal of this proposal is to better understand the basis of structural airway changes in severe asthma and how asthma exacerbations may contribute to their progression over time. The investigators propose to study a well-characterized cohort of adult and pediatric subjects with asthma using a multidisciplinary state-of-the-art approach. We hypothesize that severe asthma exacerbations, in some patients, are associated with incomplete recovery and activation of airway inflammatory cells in a regional distribution. The end result is a more permanent and less reversible airway obstruction that is a prominent feature of severe asthma.

DETAILED DESCRIPTION:
We have shown that patients with severe asthma have heterogeneous regional ventilation defects and air trapping. Some of these defects are persistent, while others can be provoked with virus-induced exacerbations or bronchial challenge and recur in the same general areas on repeated challenge, suggesting localized airway dysfunction. In preliminary studies, inflammatory parameters tended to be more prominent in segments that showed ventilation defects on imaging. Therefore, we hypothesize that asthma exacerbations, in some patients, are associated with incomplete recovery and activation of airway inflammatory cells in a regional distribution. This leads to enhanced airway injury with airway dysfunction as reflected by ventilation defects and air trapping, and a more generalized increase in disease severity. To evaluate this hypothesis we propose the following specific aims: 1. To refine phenotyping of severe asthma using new variables from multiple domains in a large longitudinal patient cohort; and to determine the contribution of asthma exacerbations to disease progression. 2. To characterize regional obstructive patterns at baseline and their relationship to changes in pulmonary function; and to determine how incremental changes in regional airway dysfunction after asthma exacerbations may contribute to severe asthma. 3. To determine the contribution of established and novel biomarkers (YKL-40, vWF, & P-selectin), in refining the severe asthma phenotypes and the role of inflammatory cells in causing airway injury following virus-induced asthma exacerbations with subsequent development of ventilation defects.

ELIGIBILITY:
Inclusion Criteria:

1. Physician diagnosis of asthma
2. Age 6 years and older
3. Evidence of historical reversibility, including either:

1. FEV1 bronchodilator reversibility ≥ 12%, or

2. Airway hyperresponsiveness reflected by a methacholine PC20 ≤16 mg/mL.

Exclusion Criteria:

1. No primary medical caregiver,
2. Pregnancy (if undergoing methacholine challenge or bronchoscopy),
3. Current smoking
4. Smoking history > 10 pack years if ≥ 30 years of age or smoking history > 5 pack years if < 30 years of age (Note: If a subject has a smoking history, no smoking within the past year)
5. Other chronic pulmonary disorders associated with asthma-like symptoms,including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal cord dysfunction that is the sole cause of asthma symptoms, severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways,
6. History of premature birth before 35 weeks gestation,
7. Evidence that the participant or family may be unreliable or poorly adherent to their asthma treatment or study procedures,
8. Planning to relocate from the clinical center area before study completion, or
9. Any other criteria that place the subject at unnecessary risk according to the judgment of the Principal Investigator and/or attending physician(s) of record.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with asthma (severe asthma, well controlled asthma) and healthy normal controls from Madison, WI region
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Lung function | Baseline versus 3 years
  Changes in airway function after a severe exacerbation, and longitudinally over 3 years, as measured by lung function.

SECONDARY OUTCOMES:
Plethysmographic lung volumes | Baseline versus 3 years
  Changes in airway function after a severe exacerbation, and longitudinally over 3 years, as measured by Plethysmographic lung volumes.
Hyperpolarized gas magnetic resonance imaging | Baseline versus 3 years
  Changes in airway function after a severe exacerbation, and longitudinally over 3 years, as measured by Hyperpolarized gas magnetic resonance imaging.
Multidetector computed tomography imaging | Baseline versus 3 years
  Changes in airway function after a severe exacerbation, and longitudinally over 3 years, as measured by Multidetector computed tomography imaging (adults only).
Exacerbations | Baseline versus 3 years
  Exacerbation requiring systemic steroids
Plasma levels of biomarkers | Baseline versus 3 years
  Changes in airway function after a severe exacerbation, and longitudinally over 3 years, as measured by plasma levels of biomarkers.
Induced sputum mediators | Baseline versus 3 years
  Changes in airway function after a severe exacerbation, and longitudinally over 3 years, as measured by induced sputum mediators.
Nasal washing samples for virology | Baseline versus 3 years
  Changes in airway function after a severe exacerbation, and longitudinally over 3 years, as measured by nasal washing samples for virology.
Bronchoscopy samples for virology, inflammatory cells and mediators | Baseline versus 3 years
  Changes in airway function after a severe exacerbation, and longitudinally over 3 years, as measured by bronchoscopy samples for virology, inflammatory cells and mediators (adults only).

CONTACTS AND LOCATIONS:
Overall Officials: Nizar N Jarjour, MD, Principal Investigator — UW Madison
Locations (1):
- UW Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang BK, Elicker BM, Henry TS, Kallianos KG, Hahn LD, Tang M, Heng F, McCulloch CE, Bhakta NR, Majumdar S, Choi J, Denlinger LC, Fain SB, Hastie AT, Hoffman EA, Israel E, Jarjour NN, Levy BD, Mauger DT, Sumino K, Wenzel SE, Castro M, Woodruff PG, Fahy JV, Sarp FTNSARP. Persistent mucus plugs in proximal airways are consequential for airflow limitation in asthma. JCI Insight. 2024 Feb 8;9(3):e174124. doi: 10.1172/jci.insight.174124. PMID 38127464
- [Derived] Dunican EM, Elicker BM, Gierada DS, Nagle SK, Schiebler ML, Newell JD, Raymond WW, Lachowicz-Scroggins ME, Di Maio S, Hoffman EA, Castro M, Fain SB, Jarjour NN, Israel E, Levy BD, Erzurum SC, Wenzel SE, Meyers DA, Bleecker ER, Phillips BR, Mauger DT, Gordon ED, Woodruff PG, Peters MC, Fahy JV; National Heart Lung and Blood Institute (NHLBI) Severe Asthma Research Program (SARP). Mucus plugs in patients with asthma linked to eosinophilia and airflow obstruction. J Clin Invest. 2018 Mar 1;128(3):997-1009. doi: 10.1172/JCI95693. Epub 2018 Feb 5. PMID 29400693
- [Derived] Denlinger LC, Phillips BR, Ramratnam S, Ross K, Bhakta NR, Cardet JC, Castro M, Peters SP, Phipatanakul W, Aujla S, Bacharier LB, Bleecker ER, Comhair SA, Coverstone A, DeBoer M, Erzurum SC, Fain SB, Fajt M, Fitzpatrick AM, Gaffin J, Gaston B, Hastie AT, Hawkins GA, Holguin F, Irani AM, Israel E, Levy BD, Ly N, Meyers DA, Moore WC, Myers R, Opina MT, Peters MC, Schiebler ML, Sorkness RL, Teague WG, Wenzel SE, Woodruff PG, Mauger DT, Fahy JV, Jarjour NN; National Heart, Lung, and Blood Institute's Severe Asthma Research Program-3 Investigators. Inflammatory and Comorbid Features of Patients with Severe Asthma and Frequent Exacerbations. Am J Respir Crit Care Med. 2017 Feb 1;195(3):302-313. doi: 10.1164/rccm.201602-0419OC. PMID 27556234
- [Derived] Witt CA, Sheshadri A, Carlstrom L, Tarsi J, Kozlowski J, Wilson B, Gierada DS, Hoffman E, Fain SB, Cook-Granroth J, Sajol G, Sierra O, Giri T, O'Neill M, Zheng J, Schechtman KB, Bacharier LB, Jarjour N, Busse W, Castro M; NHLBI Severe Asthma Research Program (SARP). Longitudinal changes in airway remodeling and air trapping in severe asthma. Acad Radiol. 2014 Aug;21(8):986-93. doi: 10.1016/j.acra.2014.05.001. PMID 25018070
- See also: SARP Website — http://severeasthma.org/